CLINICAL TRIAL: NCT00524537
Title: A Long-Term Non-Interventional Registry to Assess Safety and Effectiveness of HUMIRA® (Adalimumab) in Subjects With Moderately to Severely Active Crohn's Disease (CD)
Brief Title: A Long-Term Registry of Humira® (Adalimumab) in Subjects With Moderately to Severely Active Crohn's Disease (CD)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P06-134
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab (Humira) Treatment: Adult patients with moderately to severely active CD treated with Humira in a routine clinical practice setting.

SUMMARY:
The purpose of this Registry study is to evaluate the long-term safety and effectiveness of adalimumab in CD subjects who are treated as recommended in the product label.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are newly prescribed HUMIRA® (adalimumab) therapy (have never been treated with adalimumab) or who are participants in Abbvie sponsored investigational Crohn's disease (CD) trials, are currently receiving adalimumab and for whom the treating physician has made the decision to continue with adalimumab therapy beyond the duration of the investigational trial.
* Subjects who were participants in AbbVie sponsored investigational Crohn's CD trials, who have not had dose interruptions since the last dose of study drug, where the Investigator can provide source documentation of dosing information.
* Subjects who are currently receiving adalimumab, as per the local approved label, who have not had dose interruptions since the induction dose of adalimumab where the Investigator can provide source documentation of dosing information.
* Subjects willing to consent to data being collected and provided to AbbVie.
* Subjects capable of and willing to give written informed consent and to comply with the requirements of the Registry study protocol.

Exclusion Criteria:

- Subjects should not be enrolled if they cannot be treated in accordance with the local product label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease who have been prescribed adalimumab according to the local label.
Sampling Method: Non-Probability Sample
Enrollment: 5025 (Actual)
Dates: Start 2007-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Ahuja D, Luo J, Qi Y, Syal G, Boland BS, Chang J, Ma C, Jairath V, Xu R, Singh S. Impact of Treatment Response on Risk of Serious Infections in Patients With Crohn's Disease: Secondary Analysis of the PYRAMID Registry. Clin Gastroenterol Hepatol. 2024 Jun;22(6):1286-1294.e4. doi: 10.1016/j.cgh.2024.01.003. Epub 2024 Jan 11. PMID 38216022
- [Derived] D'Haens G, Reinisch W, Panaccione R, Satsangi J, Petersson J, Bereswill M, Arikan D, Perotti E, Robinson AM, Kalabic J, Alperovich G, Thakkar R, Loftus EV. Lymphoma Risk and Overall Safety Profile of Adalimumab in Patients With Crohn's Disease With up to 6 Years of Follow-Up in the Pyramid Registry. Am J Gastroenterol. 2018 Jun;113(6):872-882. doi: 10.1038/s41395-018-0098-4. Epub 2018 Jun 5. PMID 29867173
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 participants less than 18 years of age were enrolled in the study. Participants were permitted to re-enroll after discontinuing the study. Of the 2811 participants who discontinued study, 339 re-enrolled in the study; 102 participants discontinued from the study after re-enrollment.
Period: Overall Study
Arm/Group | Adalimumab (Humira) Treatment
Started | 5025 (All Treated Population: All participants who received at least 1 injection of Humira in the registry)
Discontinued | 2811 (Discontinued from study)
Re-enrolled | 339 (Discontinued from study and later re-enrolled in study)
Discontinued After Re-enrollment | 102 (Discontinued from study after re-enrollment)
Completed | 2451 (Still enrolled in study at the end of study)
Not Completed | 2574

BASELINE CHARACTERISTICS:
Population: All Treated Population: All participants who received at least 1 injection of Humira in the registry
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 5025
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2869
  Male | 2156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Registry Treatment-Emergent Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Registry treatment-emergent AEs are defined as any event that began or worsened in severity after the first dose of Humira in the registry. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
  For more details on adverse events please see the AE section below.
Time Frame: Registry treatment-emergent SAEs and AEs of special interest are summarized from the day of the first dose of Humira in the registry until 70 days after the last non-missing Humira injection date in the registry (up to approximately 6 years).
Population: All Treated Population: All participants who received at least 1 injection of Humira in the registry
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 5025
Participants
  Any AE | 2392
  Any SAE | 1853
  AE Leading to Discontinuation of Study Drug | 596
  Any AE Leading to Death | 43

2. Secondary Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Total Score: Change From Baseline to Each Visit
Description: The SIBDQ is a disease-specific health-related quality of life (HRQoL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) patients by measuring physical, social and emotional status. The SIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). The scores are summed up and range from 10 (poor QoL) to 70 (good QoL). A higher score indicates a better HRQoL; a positive change from baseline indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with SIBDQ measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 2166
units on a scale
  Change from Baseline to Month 12 (N=1712) | 4.98 (12.335)
  Change from Baseline to Month 24 (N=1319) | 4.20 (13.397)
  Change from Baseline to Month 36 (N=1712) | 5.01 (12.994)
  Change from Baseline to Month 48 (N=969) | 5.51 (13.466)
  Change from Baseline to Month 60 (N=837) | 5.45 (13.211)
  Change from Baseline to Month 72 (N=748) | 5.41 (12.768)

3. Secondary Outcome: Physician's Global Assessment of Disease Activity (PGA): Change From Baseline to Each Visit
Description: The PGA measures the physician's assessment of the patient's current disease activity from using 6 assessments (general well-being, abdominal pain, diarrhea, blood in stool, abdominal mass, and Crohn's disease-related complications). The PGA score is the sum of the subscores and ranges from 0 (very good) to approximately 25 (very bad). A negative change in score indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with PGA measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 3897
units on a scale
  Change from Baseline to Month 12 (N=3335) | -1.63 (4.961)
  Change from Baseline to Month 24 (N=2856) | -1.63 (5.108)
  Change from Baseline to Month 36 (N=2629) | -1.84 (5.143)
  Change from Baseline to Month 48 (N=2403) | -1.91 (5.169)
  Change from Baseline to Month 60 (N=2162) | -2.00 (5.242)
  Change from Baseline to Month 72 (N=1983) | -2.08 (5.602)

4. Secondary Outcome: Work Productivity and Activity Impairment: Special Health Problem (WPAI:SHP): Change in Mean Percentage of Work Time Missed (Absenteeism) From Baseline to Each Visit
Description: Absenteeism, presented as the mean percentage of work time missed due to Crohn's Disease (as reported on the WPAI:SHP), and is calculated as: 100*number of hours of work missed due to psoriasis / (number of hours of work missed due to psoriasis + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. A negative change in score indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with WPAI:SHP measurements.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 1065
percentage of work time missed
  Change from Baseline to Month 12 (N=829) | -4.92 (26.881)
  Change from Baseline to Month 24 (N=612) | -3.02 (26.607)
  Change from Baseline to Month 36 (N=507) | -5.62 (29.649)
  Change from Baseline to Month 48 (N=436) | -3.93 (31.884)
  Change from Baseline to Month 60 (N=368) | -3.22 (29.622)
  Change from Baseline to Month 72 (N=303) | -3.89 (26.865)

5. Secondary Outcome: WPAI:SHP: Change in Mean Percentage of Impairment While Working (Presenteeism) Due to Crohn's Disease From Baseline to Each Visit
Description: Presenteeism (the extent to which CD decreased productivity) is presented as the mean percentage of impairment while working due to CD, and is calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI:SHP is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. A negative change in score indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 1183
percentage of impairment while working
  Change from Baseline to Month 12 (N=914) | -8.00 (29.602)
  Change from Baseline to Month 24 (N=697) | -7.04 (31.666)
  Change from Baseline to Month 36 (N=577) | -9.84 (30.570)
  Change from Baseline to Month 48 (N=493) | -8.09 (33.611)
  Change from Baseline to Month 60 (N=418) | -8.21 (30.130)
  Change from Baseline to Month 72 (N=361) | -8.03 (29.472)

6. Secondary Outcome: WPAI:SHP: Change in Mean Percentage of Overall Work Impairment Due to Crohn's Disease From Baseline to Each Visit
Description: The mean percentage of overall work impairment due to CD (based on the WPAI questionnaire) is presented, and is calculated as: Absenteeism (%) + extent to which CD decreased productivity (%)* [number of hours worked / (number of hours of work missed due to CD + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. A negative change in score indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 1061
percentage of overall work impairment
  Change from Baseline to Month 12 (N=821) | -9.48 (32.976)
  Change from Baseline to Month 24 (N=605) | -7.95 (35.798)
  Change from Baseline to Month 36 (N=498) | -11.78 (34.886)
  Change from Baseline to Month 48 (N=435) | -9.15 (36.957)
  Change from Baseline to Month 60 (N=365) | -8.14 (34.696)
  Change from Baseline to Month 72 (N=300) | -9.33 (34.631)

7. Secondary Outcome: WPAI:SHP: Change in Mean Percentage of Activity Impairment Due to Crohn's Disease From Baseline to Each Visit
Description: Activity impairment due to CD (the extent to which CD affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, and is calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. A negative change in score indicates improvement. N=the number of participants with available data at both baseline and given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 2110
percentage of activity impairment
  Change from Baseline to Month 12 (N=1665) | -10.93 (30.548)
  Change from Baseline to Month 24 (N=1286) | -9.75 (33.244)
  Change from Baseline to Month 36 (N=1095) | -10.07 (32.705)
  Change from Baseline to Month 48 (N=944) | -10.14 (33.063)
  Change from Baseline to Month 60 (N=817) | -10.78 (31.787)
  Change from Baseline to Month 72 (N=718) | -11.13 (29.533)

8. Secondary Outcome: Healthcare Resource Utilization (HCRU): Mean Number Of Visits At Physician's Office Due to CD at Each Study Visit
Description: The HCRU assesses the frequency of unscheduled outpatient visits, emergency room visits, or hospitalizations for their CD in the past 3 months. The mean number of visits at physician's office in the past 3 months is presented at each timepoint. N=number of participants with at least one visit at given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with at least 1 visit at physician's office.
Measure: Mean (Standard Deviation); unit: number of visits at physician's office
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 5025
number of visits at physician's office
  Baseline (N=97) | 2.79 (2.947)
  Month 12 (N=780) | 1.95 (2.039)
  Month 24 (N=1042) | 2.19 (2.079)
  Month 36 (N=1003) | 2.38 (3.242)
  Month 48 (N=869) | 2.38 (2.326)
  Month 60 (N=798) | 2.39 (2.084)
  Month 72 (N=711) | 2.32 (2.051)

9. Secondary Outcome: Healthcare Resource Utilization (HCRU): Mean Number Of Visits At Emergency Room Due to CD at Each Study Visit
Description: The HCRU assesses the frequency of unscheduled outpatient visits, emergency room visits, or hospitalizations due to CD in the past 3 months. The mean number of visits at emergency room in the past 3 months is presented at each timepoint. N=number of participants with at least one visit at given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with at least 1 visit at emergency room.
Measure: Mean (Standard Deviation); unit: number of visits at emergency room
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 177
number of visits at emergency room
  Baseline (N=8) | 1.13 (0.354)
  Month 12 (N=143) | 1.28 (0.883)
  Month 24 (N=162) | 1.25 (0.558)
  Month 36 (N=134) | 1.49 (0.865)
  Month 48 (N=131) | 1.39 (0.686)
  Month 60 (N=124) | 1.41 (0.817)
  Month 72 (N=97) | 1.41 (0.826)

10. Secondary Outcome: Healthcare Resource Utilization (HCRU): Mean Number Of Admissions to Hospital Due to CD at Each Study Visit
Description: The HCRU assesses the frequency of unscheduled outpatient visits, emergency room visits, or hospitalizations due to CD in the past 3 months. The mean number of admissions to hospital in the past 3 months is presented at each timepoint. N=number of participants with data for "total days in hospital" and at least one admission to hospital at given timepoint..
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with data for "total days in hospital" and at least one admission to hospital.
Measure: Mean (Standard Deviation); unit: number of admissions to hospital
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 5025
number of admissions to hospital
  Baseline (N=10) | 1.30 (0.675)
  Month 12 (N=230) | 1.29 (0.780)
  Month 24 (N=255) | 1.26 (0.585)
  Month 36 (N=229) | 1.41 (0.793)
  Month 48 (N=180) | 1.54 (2.037)
  Month 60 (N=197) | 1.60 (1.215)
  Month 72 (N=180) | 1.83 (3.115)

11. Secondary Outcome: Healthcare Resource Utilization (HCRU): Mean Total Days In Hospital Due to CD at Each Study Visit
Description: The HCRU assesses the frequency of unscheduled outpatient visits, emergency room visits, or hospitalizations due to CD in the past 3 months. The mean total days in hospital in the past 3 months is presented at each timepoint. N=number of participants with data for "total days in hospital" at given timepoint.
Time Frame: Baseline (Enrollment) and 12, 24, 36, 48, 60, and 72 Months
Population: All participants in the All Treated Population (received at least 1 injection of Humira in the registry) with data for "total days in hospital".
Measure: Mean (Standard Deviation); unit: total days in hospital
Arm/Group | Adalimumab (Humira) Treatment
Number analyzed (Participants) | 260
total days in hospital
  Baseline (N=10) | 5.80 (3.259)
  Month 12 (N=230) | 8.19 (9.801)
  Month 24 (N=255) | 9.17 (11.753)
  Month 36 (N=229) | 9.75 (19.474)
  Month 48 (N=180) | 8.37 (10.011)
  Month 60 (N=195) | 9.03 (12.997)
  Month 72 (N=180) | 9.27 (13.158)

ADVERSE EVENTS:
Time Frame: Registry treatment-emergent SAEs and AEs of special interest are summarized from the day of the first dose of Humira in the registry until 70 days after the last non-missing Humira injection date in the registry (up to approximately 6 years).
Description: Treatment-emergent AEs (TEAEs) of special interest were intended to be collected; however, if TEAEs were spontaneously reported by the participant, they were also analyzed.
Arm/Group | Adalimumab (Humira) Treatment
Serious Adverse Events (participants affected / at risk) | 1853/5025
Other Adverse Events (participants affected / at risk) | 958/5025
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (Humira) Treatment (N=5025)
ANAEMIA (Blood and lymphatic system disorders) | 25
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
BONE MARROW OEDEMA (Blood and lymphatic system disorders) | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 2
EOSINOPHILIA (Blood and lymphatic system disorders) | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 2
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 3
LYMPHADENITIS (Blood and lymphatic system disorders) | 4
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 4
ANGINA PECTORIS (Cardiac disorders) | 4
ANGINA UNSTABLE (Cardiac disorders) | 2
ARTERIOSPASM CORONARY (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 4
BRADYARRHYTHMIA (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 2
CARDIAC VALVE DISEASE (Cardiac disorders) | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 3
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 8
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
PERICARDITIS (Cardiac disorders) | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
TACHYARRHYTHMIA (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 3
VENTRICULAR FIBRILLATION (Cardiac disorders) | 2
VITELLO-INTESTINAL DUCT REMNANT (Congenital, familial and genetic disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
BASEDOW'S DISEASE (Endocrine disorders) | 1
GOITRE (Endocrine disorders) | 2
BLEPHARITIS (Eye disorders) | 1
CORNEAL DISORDER (Eye disorders) | 1
EPISCLERITIS (Eye disorders) | 1
RETINOPATHY (Eye disorders) | 1
SCLERITIS (Eye disorders) | 1
ULCERATIVE KERATITIS (Eye disorders) | 1
VISUAL IMPAIRMENT (Eye disorders) | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 12
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
ABDOMINAL HERNIA (Gastrointestinal disorders) | 10
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1
ABDOMINAL MASS (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 61
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8
ABDOMINAL WALL DISORDER (Gastrointestinal disorders) | 1
ABNORMAL FAECES (Gastrointestinal disorders) | 1
ANAL FISSURE (Gastrointestinal disorders) | 7
ANAL FISTULA (Gastrointestinal disorders) | 84
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ANAL SPHINCTER ATONY (Gastrointestinal disorders) | 1
ANAL STENOSIS (Gastrointestinal disorders) | 12
ANAL ULCER (Gastrointestinal disorders) | 1
ANOGENITAL DYSPLASIA (Gastrointestinal disorders) | 1
ANORECTAL DISORDER (Gastrointestinal disorders) | 8
ANORECTAL STENOSIS (Gastrointestinal disorders) | 2
APHTHOUS ULCER (Gastrointestinal disorders) | 2
ASCITES (Gastrointestinal disorders) | 4
AUTOIMMUNE PANCREATITIS (Gastrointestinal disorders) | 1
COELIAC ARTERY COMPRESSION SYNDROME (Gastrointestinal disorders) | 1
COLITIS (Gastrointestinal disorders) | 17
COLITIS ULCERATIVE (Gastrointestinal disorders) | 4
COLON DYSPLASIA (Gastrointestinal disorders) | 4
COLONIC FISTULA (Gastrointestinal disorders) | 8
CONSTIPATION (Gastrointestinal disorders) | 13
CROHN'S DISEASE (Gastrointestinal disorders) | 606
DEFAECATION URGENCY (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 24
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
DIEULAFOY'S VASCULAR MALFORMATION (Gastrointestinal disorders) | 1
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 2
DUODENAL STENOSIS (Gastrointestinal disorders) | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 2
ENTERITIS (Gastrointestinal disorders) | 15
ENTEROCOLONIC FISTULA (Gastrointestinal disorders) | 7
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 22
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 5
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1
FAECAL INCONTINENCE (Gastrointestinal disorders) | 2
FAECALOMA (Gastrointestinal disorders) | 2
FAECES DISCOLOURED (Gastrointestinal disorders) | 2
FEMORAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 7
FOOD POISONING (Gastrointestinal disorders) | 2
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 2
GASTRIC FISTULA (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 5
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 2
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 1
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 4
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 3
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL STENOSIS (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3
HAEMATEMESIS (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 2
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1
ILEAL PERFORATION (Gastrointestinal disorders) | 1
ILEAL STENOSIS (Gastrointestinal disorders) | 94
ILEUS (Gastrointestinal disorders) | 13
ILEUS PARALYTIC (Gastrointestinal disorders) | 2
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 4
INFREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 2
INTERNAL HERNIA (Gastrointestinal disorders) | 1
INTESTINAL DILATATION (Gastrointestinal disorders) | 2
INTESTINAL FIBROSIS (Gastrointestinal disorders) | 1
INTESTINAL FISTULA (Gastrointestinal disorders) | 12
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1
INTESTINAL MASS (Gastrointestinal disorders) | 1
INTESTINAL MUCOSAL HYPERTROPHY (Gastrointestinal disorders) | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 127
INTESTINAL PERFORATION (Gastrointestinal disorders) | 8
INTESTINAL POLYP (Gastrointestinal disorders) | 1
INTESTINAL STENOSIS (Gastrointestinal disorders) | 44
INTESTINAL ULCER (Gastrointestinal disorders) | 1
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 2
INTUSSUSCEPTION (Gastrointestinal disorders) | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 2
JEJUNAL PERFORATION (Gastrointestinal disorders) | 2
JEJUNAL STENOSIS (Gastrointestinal disorders) | 6
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 12
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 41
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 6
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 2
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2
MEGACOLON (Gastrointestinal disorders) | 3
MELAENA (Gastrointestinal disorders) | 1
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 3
NARCOTIC BOWEL SYNDROME (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 16
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 1
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 1
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 2
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 2
OESOPHAGITIS (Gastrointestinal disorders) | 2
OMENTAL INFARCTION (Gastrointestinal disorders) | 1
ORAL DISORDER (Gastrointestinal disorders) | 1
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 7
PANCREATITIS ACUTE (Gastrointestinal disorders) | 8
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 1
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 1
PAPILLA OF VATER STENOSIS (Gastrointestinal disorders) | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1
PHARYNGO-OESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 1
POUCHITIS (Gastrointestinal disorders) | 2
PROCTALGIA (Gastrointestinal disorders) | 8
PROCTITIS (Gastrointestinal disorders) | 6
PSEUDOPOLYPOSIS (Gastrointestinal disorders) | 1
RECTAL DISCHARGE (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 14
RECTAL PERFORATION (Gastrointestinal disorders) | 1
RECTAL SPASM (Gastrointestinal disorders) | 1
RECTAL STENOSIS (Gastrointestinal disorders) | 8
SHORT-BOWEL SYNDROME (Gastrointestinal disorders) | 2
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 131
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 5
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 21
SMALL INTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 68
TOOTHACHE (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3
VOLVULUS OF SMALL BOWEL (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 18
ASTHENIA (General disorders) | 8
CATHETER SITE DISCHARGE (General disorders) | 1
CHEST PAIN (General disorders) | 2
CHILLS (General disorders) | 4
CYST (General disorders) | 1
DEATH (General disorders) | 2
DEVICE DISLOCATION (General disorders) | 1
DEVICE ISSUE (General disorders) | 1
DEVICE LEAKAGE (General disorders) | 1
DISCOMFORT (General disorders) | 1
DRUG EFFECT DECREASED (General disorders) | 2
DRUG INTOLERANCE (General disorders) | 3
DRUG WITHDRAWAL SYNDROME (General disorders) | 1
DYSPLASIA (General disorders) | 1
FACE OEDEMA (General disorders) | 1
FIBROSIS (General disorders) | 1
GAIT DISTURBANCE (General disorders) | 3
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 7
HYPERTHERMIA (General disorders) | 1
IMPAIRED HEALING (General disorders) | 5
INFLAMMATION (General disorders) | 1
LOCAL SWELLING (General disorders) | 1
LOCALISED OEDEMA (General disorders) | 1
MALAISE (General disorders) | 4
MASS (General disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 3
NO THERAPEUTIC RESPONSE (General disorders) | 4
NON-CARDIAC CHEST PAIN (General disorders) | 3
OEDEMA (General disorders) | 3
OEDEMA PERIPHERAL (General disorders) | 3
PAIN (General disorders) | 2
PYREXIA (General disorders) | 27
SENSATION OF FOREIGN BODY (General disorders) | 1
SUDDEN DEATH (General disorders) | 2
TREATMENT FAILURE (General disorders) | 1
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1
BILE DUCT STONE (Hepatobiliary disorders) | 2
BILIARY COLIC (Hepatobiliary disorders) | 5
CHOLANGITIS (Hepatobiliary disorders) | 5
CHOLANGITIS CHRONIC (Hepatobiliary disorders) | 1
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 5
CHOLECYSTITIS (Hepatobiliary disorders) | 9
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 18
CHOLELITHIASIS OBSTRUCTIVE (Hepatobiliary disorders) | 1
CIRRHOSIS ALCOHOLIC (Hepatobiliary disorders) | 1
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1
HEPATIC NECROSIS (Hepatobiliary disorders) | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 1
HEPATITIS ALCOHOLIC (Hepatobiliary disorders) | 1
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1
JAUNDICE (Hepatobiliary disorders) | 1
NODULAR REGENERATIVE HYPERPLASIA (Hepatobiliary disorders) | 1
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 2
AMYLOIDOSIS (Immune system disorders) | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 3
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 2
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 1
TRANSPLANT REJECTION (Immune system disorders) | 1
ABDOMINAL ABSCESS (Infections and infestations) | 43
ABDOMINAL INFECTION (Infections and infestations) | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 3
ABSCESS (Infections and infestations) | 18
ABSCESS INTESTINAL (Infections and infestations) | 19
ABSCESS JAW (Infections and infestations) | 1
ABSCESS LIMB (Infections and infestations) | 2
ACUTE SINUSITIS (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 119
ANAL FISTULA INFECTION (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 7
APPENDICITIS PERFORATED (Infections and infestations) | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 2
BACTERAEMIA (Infections and infestations) | 3
BARTHOLIN'S ABSCESS (Infections and infestations) | 1
BARTHOLINITIS (Infections and infestations) | 1
BILIARY SEPSIS (Infections and infestations) | 1
BRAIN ABSCESS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 6
BRONCHITIS BACTERIAL (Infections and infestations) | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 4
CAMPYLOBACTER INFECTION (Infections and infestations) | 2
CANDIDA INFECTION (Infections and infestations) | 2
CANDIDA PNEUMONIA (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 19
CHOLANGITIS INFECTIVE (Infections and infestations) | 1
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 3
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 8
CYSTITIS (Infections and infestations) | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 5
DEVICE RELATED SEPSIS (Infections and infestations) | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 2
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 3
EAR INFECTION (Infections and infestations) | 2
ENDOCARDITIS (Infections and infestations) | 3
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 4
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1
ESCHERICHIA INFECTION (Infections and infestations) | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 2
FALLOPIAN TUBE ABSCESS (Infections and infestations) | 1
FUNGAEMIA (Infections and infestations) | 1
FUNGAL PERITONITIS (Infections and infestations) | 1
GAS GANGRENE (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 26
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 5
GASTROINTESTINAL INFECTION (Infections and infestations) | 4
GENITAL ABSCESS (Infections and infestations) | 3
GENITAL HERPES (Infections and infestations) | 1
GENITAL INFECTION (Infections and infestations) | 1
GROIN ABSCESS (Infections and infestations) | 5
H1N1 INFLUENZA (Infections and infestations) | 2
HAEMATOMA INFECTION (Infections and infestations) | 1
HAEMOPHILUS INFECTION (Infections and infestations) | 1
HELICOBACTER GASTRITIS (Infections and infestations) | 1
HELICOBACTER INFECTION (Infections and infestations) | 1
HEPATITIS C (Infections and infestations) | 1
HERPES OESOPHAGITIS (Infections and infestations) | 1
HERPES OPHTHALMIC (Infections and infestations) | 1
HERPES SIMPLEX (Infections and infestations) | 2
HERPES VIRUS INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 8
HERPES ZOSTER OTICUS (Infections and infestations) | 2
HIV INFECTION (Infections and infestations) | 1
IMPETIGO (Infections and infestations) | 1
INCISION SITE ABSCESS (Infections and infestations) | 2
INFECTED CYST (Infections and infestations) | 2
INFECTION (Infections and infestations) | 3
INFECTION PARASITIC (Infections and infestations) | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 5
INTERVERTEBRAL DISCITIS (Infections and infestations) | 2
KIDNEY INFECTION (Infections and infestations) | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1
LEGIONELLA INFECTION (Infections and infestations) | 1
LISTERIOSIS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
LUNG ABSCESS (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 1
LYMPHADENITIS BACTERIAL (Infections and infestations) | 1
MASTITIS (Infections and infestations) | 1
MASTOIDITIS (Infections and infestations) | 1
MENINGITIS VIRAL (Infections and infestations) | 1
MUSCLE ABSCESS (Infections and infestations) | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 2
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 4
OPHTHALMIC HERPES SIMPLEX (Infections and infestations) | 1
ORAL CANDIDIASIS (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 2
ORCHITIS (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 2
OTITIS EXTERNA (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 3
OVERGROWTH BACTERIAL (Infections and infestations) | 2
PAROTITIS (Infections and infestations) | 1
PELVIC ABSCESS (Infections and infestations) | 13
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1
PERINEAL ABSCESS (Infections and infestations) | 6
PERIORBITAL CELLULITIS (Infections and infestations) | 1
PERIRECTAL ABSCESS (Infections and infestations) | 14
PERITONEAL ABSCESS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 16
PERITONITIS BACTERIAL (Infections and infestations) | 1
PERIUMBILICAL ABSCESS (Infections and infestations) | 1
PERTUSSIS (Infections and infestations) | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 2
PILONIDAL CYST (Infections and infestations) | 6
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 3
PNEUMONIA (Infections and infestations) | 33
PNEUMONIA BACTERIAL (Infections and infestations) | 2
PNEUMONIA CHLAMYDIAL (Infections and infestations) | 1
PNEUMONIA FUNGAL (Infections and infestations) | 1
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 2
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 1
POST PROCEDURAL SEPSIS (Infections and infestations) | 2
POSTOPERATIVE ABSCESS (Infections and infestations) | 5
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 10
PSOAS ABSCESS (Infections and infestations) | 5
PULMONARY TUBERCULOSIS (Infections and infestations) | 5
PYELONEPHRITIS (Infections and infestations) | 4
PYELONEPHRITIS ACUTE (Infections and infestations) | 4
RECTAL ABSCESS (Infections and infestations) | 21
RENAL ABSCESS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1
RETROPERITONEAL ABSCESS (Infections and infestations) | 2
RICKETTSIOSIS (Infections and infestations) | 1
SALMONELLOSIS (Infections and infestations) | 2
SALPINGITIS (Infections and infestations) | 1
SCROTAL ABSCESS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 19
SEPTIC SHOCK (Infections and infestations) | 5
SIALOADENITIS (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 4
SKIN CANDIDA (Infections and infestations) | 1
SOFT TISSUE INFECTION (Infections and infestations) | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 9
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2
STOMA SITE ABSCESS (Infections and infestations) | 3
STREPTOCOCCAL INFECTION (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 12
SUBDIAPHRAGMATIC ABSCESS (Infections and infestations) | 1
SUPERINFECTION BACTERIAL (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 3
TOOTH ABSCESS (Infections and infestations) | 1
TORULOPSIS INFECTION (Infections and infestations) | 1
TRACHEITIS (Infections and infestations) | 1
TRACHEOBRONCHITIS (Infections and infestations) | 1
TUBERCULOSIS (Infections and infestations) | 3
TUBERCULOSIS GASTROINTESTINAL (Infections and infestations) | 1
TUBO-OVARIAN ABSCESS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 14
UROSEPSIS (Infections and infestations) | 4
VAGINAL ABSCESS (Infections and infestations) | 1
VARICELLA (Infections and infestations) | 1
VARICELLA ZOSTER PNEUMONIA (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 4
VIRAL PHARYNGITIS (Infections and infestations) | 1
VULVAL ABSCESS (Infections and infestations) | 4
VULVAL CELLULITIS (Infections and infestations) | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 2
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC FISTULA (Injury, poisoning and procedural complications) | 5
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 4
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 12
ANASTOMOTIC ULCER (Injury, poisoning and procedural complications) | 2
ANASTOMOTIC ULCER HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1
COLON INJURY (Injury, poisoning and procedural complications) | 1
COMPLICATIONS OF TRANSPLANTED KIDNEY (Injury, poisoning and procedural complications) | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 2
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 4
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL DISORDER POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 16
HEAD INJURY (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 11
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 23
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
LACERATION (Injury, poisoning and procedural complications) | 2
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1
NERVE INJURY (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 4
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 7
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 2
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 4
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 3
SCAR (Injury, poisoning and procedural complications) | 1
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1
STOMA SITE INFLAMMATION (Injury, poisoning and procedural complications) | 1
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 5
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 3
UTERINE RUPTURE (Injury, poisoning and procedural complications) | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
WOUND DECOMPOSITION (Injury, poisoning and procedural complications) | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2
WOUND SECRETION (Injury, poisoning and procedural complications) | 3
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1
BACTERIAL TEST POSITIVE (Investigations) | 1
CLOSTRIDIUM TEST POSITIVE (Investigations) | 1
CSF CULTURE POSITIVE (Investigations) | 1
CULTURE URINE (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2
OXYGEN SATURATION DECREASED (Investigations) | 1
PROTEIN TOTAL ABNORMAL (Investigations) | 1
WEIGHT DECREASED (Investigations) | 5
CACHEXIA (Metabolism and nutrition disorders) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 4
DEHYDRATION (Metabolism and nutrition disorders) | 13
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 12
OBESITY (Metabolism and nutrition disorders) | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 5
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 2
FISTULA (Musculoskeletal and connective tissue disorders) | 22
FISTULA DISCHARGE (Musculoskeletal and connective tissue disorders) | 21
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 3
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 6
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
POLYCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
SERONEGATIVE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1
ACROCHORDON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
ADENOID CYSTIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
BLADDER CANCER STAGE I, WITHOUT CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CARCINOID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
CARCINOID TUMOUR OF THE APPENDIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
COLON CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
FOLLICLE CENTRE LYMPHOMA, FOLLICULAR GRADE I, II, III STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GALLBLADDER ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GALLBLADDER CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
INTRADUCTAL PAPILLOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INTRAOCULAR MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MYCOSIS FUNGOIDES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
SEMINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SMALL INTESTINE ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF THE VULVA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
VULVAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ARACHNOIDITIS (Nervous system disorders) | 1
ATAXIA (Nervous system disorders) | 1
CAROTID ARTERY ANEURYSM (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 2
CEREBRAL ARTERY EMBOLISM (Nervous system disorders) | 1
CEREBRAL CYST (Nervous system disorders) | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1
DEMYELINATION (Nervous system disorders) | 2
DIZZINESS (Nervous system disorders) | 1
DYSARTHRIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
EPILEPSY (Nervous system disorders) | 2
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 3
HEMIPARESIS (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 2
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 3
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 2
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3
OPTIC NEURITIS (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 3
POLYNEUROPATHY (Nervous system disorders) | 2
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 2
SEIZURE (Nervous system disorders) | 3
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2
SYNCOPE (Nervous system disorders) | 3
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1
UPPER MOTOR NEURONE LESION (Nervous system disorders) | 1
VIITH NERVE PARALYSIS (Nervous system disorders) | 3
ABORTION (Pregnancy, puerperium and perinatal conditions) | 4
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 23
ABORTION SPONTANEOUS COMPLETE (Pregnancy, puerperium and perinatal conditions) | 1
COMPLICATION OF DELIVERY (Pregnancy, puerperium and perinatal conditions) | 1
DELAYED DELIVERY (Pregnancy, puerperium and perinatal conditions) | 1
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 6
FOETAL DEATH (Pregnancy, puerperium and perinatal conditions) | 2
HYDROPS FOETALIS (Pregnancy, puerperium and perinatal conditions) | 1
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 3
PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 1
PROLONGED PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1
RUPTURED ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 1
AFFECTIVE DISORDER (Psychiatric disorders) | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1
COMPLETED SUICIDE (Psychiatric disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 6
DRUG DEPENDENCE (Psychiatric disorders) | 3
EATING DISORDER (Psychiatric disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 14
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1
CALCULUS URETERIC (Renal and urinary disorders) | 4
CALCULUS URINARY (Renal and urinary disorders) | 4
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
GLOMERULONEPHRITIS (Renal and urinary disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 5
NEPHROLITHIASIS (Renal and urinary disorders) | 25
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 1
PELVI-URETERIC OBSTRUCTION (Renal and urinary disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 9
RENAL FAILURE (Renal and urinary disorders) | 9
RENAL IMPAIRMENT (Renal and urinary disorders) | 2
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1
URETERIC OBSTRUCTION (Renal and urinary disorders) | 3
URETERIC STENOSIS (Renal and urinary disorders) | 1
URGE INCONTINENCE (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 3
BARTHOLIN'S CYST (Reproductive system and breast disorders) | 1
BREAST DYSPLASIA (Reproductive system and breast disorders) | 1
BREAST HYPERPLASIA (Reproductive system and breast disorders) | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1
CERVIX DISORDER (Reproductive system and breast disorders) | 1
CERVIX INFLAMMATION (Reproductive system and breast disorders) | 1
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1
ENDOMETRIAL THICKENING (Reproductive system and breast disorders) | 1
ENDOMETRIOSIS (Reproductive system and breast disorders) | 4
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 22
GENITAL PAIN (Reproductive system and breast disorders) | 1
INFERTILITY (Reproductive system and breast disorders) | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1
METRORRHAGIA (Reproductive system and breast disorders) | 1
OEDEMA GENITAL (Reproductive system and breast disorders) | 1
OVARIAN CYST (Reproductive system and breast disorders) | 5
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 1
PELVIC ADHESIONS (Reproductive system and breast disorders) | 1
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 1
PERINEAL FISTULA (Reproductive system and breast disorders) | 5
PERINEAL PAIN (Reproductive system and breast disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1
VAGINAL DISORDER (Reproductive system and breast disorders) | 1
VAGINAL FISTULA (Reproductive system and breast disorders) | 1
VARICOCELE (Reproductive system and breast disorders) | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 3
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3
BRONCHOLITHIASIS (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL TURBINATE ABNORMALITY (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 4
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 6
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 13
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY SARCOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
BLISTER (Skin and subcutaneous tissue disorders) | 1
CUTANEOUS LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 1
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 1
DERMATOSIS (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 3
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1
GUTTATE PSORIASIS (Skin and subcutaneous tissue disorders) | 1
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 2
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 4
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 3
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 3
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 4
RASH FOLLICULAR (Skin and subcutaneous tissue disorders) | 1
ABORTION INDUCED (Surgical and medical procedures) | 11
COLOSTOMY (Surgical and medical procedures) | 1
DRUG DETOXIFICATION (Surgical and medical procedures) | 1
HYSTERECTOMY (Surgical and medical procedures) | 1
INTESTINAL ANASTOMOSIS (Surgical and medical procedures) | 1
AORTIC ANEURYSM (Vascular disorders) | 1
AORTIC DISSECTION (Vascular disorders) | 1
AORTIC THROMBOSIS (Vascular disorders) | 1
ARTERIAL THROMBOSIS (Vascular disorders) | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1
BEHCET'S SYNDROME (Vascular disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 13
EMBOLISM (Vascular disorders) | 1
HAEMORRHAGE (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 2
HYPOTENSION (Vascular disorders) | 4
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2
PERIPHERAL EMBOLISM (Vascular disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
PHLEBITIS (Vascular disorders) | 1
POLYARTERITIS NODOSA (Vascular disorders) | 1
SHOCK HAEMORRHAGIC (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
VASCULITIS (Vascular disorders) | 1
VENA CAVA THROMBOSIS (Vascular disorders) | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (Humira) Treatment (N=5025)
ABDOMINAL LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 30
HYPERGAMMAGLOBULINAEMIA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 16
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 1
MACROCYTOSIS (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
SPLENIC VEIN THROMBOSIS (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3
EXTRASYSTOLES (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 2
TACHYARRHYTHMIA (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
HEREDITARY FRUCTOSE INTOLERANCE (Congenital, familial and genetic disorders) | 1
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1
EAR PAIN (Ear and labyrinth disorders) | 2
HYPOACUSIS (Ear and labyrinth disorders) | 2
TINNITUS (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 3
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1
BASEDOW'S DISEASE (Endocrine disorders) | 1
HYPERPARATHYROIDISM (Endocrine disorders) | 1
HYPOTHYROIDISM (Endocrine disorders) | 2
BLEPHARITIS (Eye disorders) | 1
CHALAZION (Eye disorders) | 1
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 2
DRY EYE (Eye disorders) | 2
EPISCLERITIS (Eye disorders) | 1
EYE INFLAMMATION (Eye disorders) | 1
IRIDOCYCLITIS (Eye disorders) | 1
IRITIS (Eye disorders) | 2
PUNCTATE KERATITIS (Eye disorders) | 1
SCLERITIS (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 2
VISUAL ACUITY REDUCED (Eye disorders) | 1
VISUAL IMPAIRMENT (Eye disorders) | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3
ABDOMINAL MASS (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 30
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 12
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1
ANAL FISSURE (Gastrointestinal disorders) | 4
ANAL FISTULA (Gastrointestinal disorders) | 13
ANAL INFLAMMATION (Gastrointestinal disorders) | 1
ANAL PRURITUS (Gastrointestinal disorders) | 2
ANAL STENOSIS (Gastrointestinal disorders) | 3
ANAL ULCER (Gastrointestinal disorders) | 1
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 1
ANORECTAL DISORDER (Gastrointestinal disorders) | 1
ANORECTAL STENOSIS (Gastrointestinal disorders) | 1
ANORECTAL SWELLING (Gastrointestinal disorders) | 1
APHTHOUS ULCER (Gastrointestinal disorders) | 3
CHAPPED LIPS (Gastrointestinal disorders) | 1
CHEILITIS GRANULOMATOSA (Gastrointestinal disorders) | 1
COELIAC DISEASE (Gastrointestinal disorders) | 1
COLITIS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 11
CROHN'S DISEASE (Gastrointestinal disorders) | 81
DENTAL CARIES (Gastrointestinal disorders) | 1
DENTAL DISCOMFORT (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 26
DIVERTICULUM (Gastrointestinal disorders) | 1
DRY MOUTH (Gastrointestinal disorders) | 1
DUODENAL STENOSIS (Gastrointestinal disorders) | 1
DUODENITIS (Gastrointestinal disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 11
DYSPHAGIA (Gastrointestinal disorders) | 2
ENTERITIS (Gastrointestinal disorders) | 2
ENTEROCOLONIC FISTULA (Gastrointestinal disorders) | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 2
FAECAL INCONTINENCE (Gastrointestinal disorders) | 4
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 2
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 2
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 4
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1
GLOSSITIS (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 3
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 5
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1
ILEAL STENOSIS (Gastrointestinal disorders) | 11
INGUINAL HERNIA (Gastrointestinal disorders) | 4
INTESTINAL FISTULA (Gastrointestinal disorders) | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
INTESTINAL STENOSIS (Gastrointestinal disorders) | 2
JEJUNAL ULCER (Gastrointestinal disorders) | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 3
LIP SWELLING (Gastrointestinal disorders) | 2
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1
MUCOUS STOOLS (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 9
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 1
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 1
ORAL LICHEN PLANUS (Gastrointestinal disorders) | 1
ORAL MUCOSAL ERUPTION (Gastrointestinal disorders) | 1
PALATAL DYSPLASIA (Gastrointestinal disorders) | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1
PERIANAL ERYTHEMA (Gastrointestinal disorders) | 2
PROCTALGIA (Gastrointestinal disorders) | 5
PROCTITIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3
RECTAL LESION (Gastrointestinal disorders) | 1
RECTAL STENOSIS (Gastrointestinal disorders) | 4
RECTAL TENESMUS (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 2
STOMATITIS (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 3
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 1
TOOTH LOSS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 9
ADVERSE DRUG REACTION (General disorders) | 1
APPLICATION SITE PAIN (General disorders) | 1
ASTHENIA (General disorders) | 7
CHEST PAIN (General disorders) | 2
CYST (General disorders) | 1
DRUG EFFECT DECREASED (General disorders) | 1
DRUG INEFFECTIVE (General disorders) | 1
DRUG INTOLERANCE (General disorders) | 4
FATIGUE (General disorders) | 7
FEELING ABNORMAL (General disorders) | 1
FEELING COLD (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
GRANULOMA (General disorders) | 1
HERNIA (General disorders) | 1
INFLAMMATION (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 7
INJECTION SITE ERYTHEMA (General disorders) | 5
INJECTION SITE INDURATION (General disorders) | 2
INJECTION SITE INFLAMMATION (General disorders) | 1
INJECTION SITE IRRITATION (General disorders) | 1
INJECTION SITE OEDEMA (General disorders) | 1
INJECTION SITE PRURITUS (General disorders) | 3
INJECTION SITE RASH (General disorders) | 1
INJECTION SITE REACTION (General disorders) | 2
INJECTION SITE SWELLING (General disorders) | 3
INJECTION SITE WARMTH (General disorders) | 1
LOCALISED OEDEMA (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 4
PAIN (General disorders) | 3
PARADOXICAL DRUG REACTION (General disorders) | 1
PERIPHERAL SWELLING (General disorders) | 2
PUNCTURE SITE REACTION (General disorders) | 1
PYREXIA (General disorders) | 17
XEROSIS (General disorders) | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 3
CHOLESTASIS (Hepatobiliary disorders) | 1
FATTY LIVER ALCOHOLIC (Hepatobiliary disorders) | 1
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1
HEPATIC CYST (Hepatobiliary disorders) | 1
HEPATIC FIBROSIS (Hepatobiliary disorders) | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
HEPATITIS (Hepatobiliary disorders) | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 1
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1
HEPATOSPLENOMEGALY (Hepatobiliary disorders) | 1
LIVER INJURY (Hepatobiliary disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 3
HYPERSENSITIVITY (Immune system disorders) | 3
SEASONAL ALLERGY (Immune system disorders) | 3
SERUM SICKNESS (Immune system disorders) | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1
ABDOMINAL WALL INFECTION (Infections and infestations) | 1
ABSCESS (Infections and infestations) | 3
ABSCESS LIMB (Infections and infestations) | 1
ACUTE SINUSITIS (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 14
ANAL INFECTION (Infections and infestations) | 1
ANGULAR CHEILITIS (Infections and infestations) | 1
BACTERIAL INFECTION (Infections and infestations) | 2
BARTHOLIN'S ABSCESS (Infections and infestations) | 2
BARTHOLINITIS (Infections and infestations) | 3
BODY TINEA (Infections and infestations) | 2
BORRELIA INFECTION (Infections and infestations) | 2
BRONCHITIS (Infections and infestations) | 18
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1
CAMPYLOBACTER INFECTION (Infections and infestations) | 1
CANDIDA INFECTION (Infections and infestations) | 8
CELLULITIS (Infections and infestations) | 8
CHLAMYDIAL INFECTION (Infections and infestations) | 1
CHRONIC HEPATITIS C (Infections and infestations) | 1
CHRONIC SINUSITIS (Infections and infestations) | 2
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 5
CONJUNCTIVITIS (Infections and infestations) | 4
CRYPTOCOCCOSIS (Infections and infestations) | 1
CRYPTOSPORIDIOSIS INFECTION (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 6
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 4
DERMO-HYPODERMITIS (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
EAR INFECTION (Infections and infestations) | 5
ECZEMA INFECTED (Infections and infestations) | 1
ENTEROBIASIS (Infections and infestations) | 1
ENTEROCOCCAL INFECTION (Infections and infestations) | 1
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 2
EYE INFECTION (Infections and infestations) | 1
EYE INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1
FOLLICULITIS (Infections and infestations) | 11
FUNGAL INFECTION (Infections and infestations) | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 2
GASTROENTERITIS (Infections and infestations) | 12
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 1
GENITAL CANDIDIASIS (Infections and infestations) | 1
GENITAL HERPES (Infections and infestations) | 3
GENITAL INFECTION FUNGAL (Infections and infestations) | 1
GINGIVAL ABSCESS (Infections and infestations) | 1
GROIN ABSCESS (Infections and infestations) | 2
GYNAECOLOGICAL CHLAMYDIA INFECTION (Infections and infestations) | 1
HERPES OPHTHALMIC (Infections and infestations) | 2
HERPES SIMPLEX (Infections and infestations) | 2
HERPES VIRUS INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 48
HIV INFECTION (Infections and infestations) | 1
INCISION SITE ABSCESS (Infections and infestations) | 2
INFECTION (Infections and infestations) | 1
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 17
INFUSION SITE INFECTION (Infections and infestations) | 1
LARYNGITIS (Infections and infestations) | 6
LATENT TUBERCULOSIS (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11
LUNG INFECTION (Infections and infestations) | 1
MASTITIS (Infections and infestations) | 2
MASTOIDITIS (Infections and infestations) | 1
MOLLUSCUM CONTAGIOSUM (Infections and infestations) | 1
MYCOBACTERIUM MARINUM INFECTION (Infections and infestations) | 1
NAIL CANDIDA (Infections and infestations) | 1
NASAL ABSCESS (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 45
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 6
ONYCHOMYCOSIS (Infections and infestations) | 1
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 2
ORAL CANDIDIASIS (Infections and infestations) | 7
ORAL FUNGAL INFECTION (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 12
ORAL INFECTION (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
OTITIS EXTERNA (Infections and infestations) | 4
OTITIS MEDIA (Infections and infestations) | 2
OVERGROWTH BACTERIAL (Infections and infestations) | 1
PAPILLOMA VIRAL INFECTION (Infections and infestations) | 2
PARONYCHIA (Infections and infestations) | 1
PAROTITIS (Infections and infestations) | 1
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1
PERIODONTITIS (Infections and infestations) | 1
PERIRECTAL ABSCESS (Infections and infestations) | 2
PHARYNGITIS (Infections and infestations) | 3
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1
PILONIDAL CYST (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 18
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2
PSEUDOMONAS INFECTION (Infections and infestations) | 1
PURULENT DISCHARGE (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 1
RASH PUSTULAR (Infections and infestations) | 1
RECTAL ABSCESS (Infections and infestations) | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 2
SALPINGITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
SIALOADENITIS (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 13
SKIN BACTERIAL INFECTION (Infections and infestations) | 1
SKIN CANDIDA (Infections and infestations) | 1
SKIN INFECTION (Infections and infestations) | 4
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 3
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1
STOMA SITE ABSCESS (Infections and infestations) | 1
STOMA SITE CANDIDA (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 7
SUPERINFECTION (Infections and infestations) | 1
TINEA PEDIS (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 8
TOOTH ABSCESS (Infections and infestations) | 3
TOOTH INFECTION (Infections and infestations) | 2
TRICHOPHYTOSIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11
UREAPLASMA INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 33
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1
UTERINE INFECTION (Infections and infestations) | 1
VAGINAL ABSCESS (Infections and infestations) | 2
VAGINAL INFECTION (Infections and infestations) | 2
VARICELLA (Infections and infestations) | 2
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 6
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 4
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 4
WOUND INFECTION (Infections and infestations) | 1
ACCIDENT AT HOME (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 4
ANASTOMOTIC ULCER (Injury, poisoning and procedural complications) | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2
FOREIGN BODY (Injury, poisoning and procedural complications) | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 3
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2
LIMB INJURY (Injury, poisoning and procedural complications) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL INFLAMMATION (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SEROMA (Injury, poisoning and procedural complications) | 1
STOMA SITE PAIN (Injury, poisoning and procedural complications) | 2
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 1
WOUND SECRETION (Injury, poisoning and procedural complications) | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ALPHA 1 FOETOPROTEIN INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 4
BLOOD IRON DECREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 2
CRYSTAL URINE (Investigations) | 1
DOUBLE STRANDED DNA ANTIBODY POSITIVE (Investigations) | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1
GIARDIA TEST POSITIVE (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HUMAN PAPILLOMA VIRUS TEST POSITIVE (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 3
RED BLOOD CELLS URINE (Investigations) | 1
SERUM FERRITIN DECREASED (Investigations) | 2
STOOL TRYPSIN (Investigations) | 1
TUBERCULIN TEST POSITIVE (Investigations) | 3
VITAMIN B12 DECREASED (Investigations) | 2
WEIGHT DECREASED (Investigations) | 4
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 6
HAEMOCHROMATOSIS (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 5
LATENT AUTOIMMUNE DIABETES IN ADULTS (Metabolism and nutrition disorders) | 1
POLYDIPSIA (Metabolism and nutrition disorders) | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 3
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 38
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1
FISTULA (Musculoskeletal and connective tissue disorders) | 7
FISTULA DISCHARGE (Musculoskeletal and connective tissue disorders) | 9
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 11
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 7
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4
OSTEITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 4
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 2
SPINAL DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 9
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 4
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 2
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CARCINOMA IN SITU OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PENILE WART (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 1
BURNING SENSATION (Nervous system disorders) | 1
CLUSTER HEADACHE (Nervous system disorders) | 1
DEMYELINATION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 2
DIZZINESS POSTURAL (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
EPILEPSY (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 22
LETHARGY (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 4
MIGRAINE WITH AURA (Nervous system disorders) | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 4
PARAESTHESIA (Nervous system disorders) | 7
SCIATICA (Nervous system disorders) | 1
SEIZURE (Nervous system disorders) | 1
SPEECH DISORDER (Nervous system disorders) | 1
TEMPORAL LOBE EPILEPSY (Nervous system disorders) | 1
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1
VIITH NERVE PARALYSIS (Nervous system disorders) | 3
UTERINE CONTRACTIONS DURING PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1
AGITATION (Psychiatric disorders) | 1
ANTICIPATORY ANXIETY (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 17
INSOMNIA (Psychiatric disorders) | 6
MENTAL DISORDER (Psychiatric disorders) | 1
PANIC REACTION (Psychiatric disorders) | 1
SLEEP DISORDER (Psychiatric disorders) | 2
STRESS (Psychiatric disorders) | 1
BLADDER SPASM (Renal and urinary disorders) | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2
DYSURIA (Renal and urinary disorders) | 1
IGA NEPHROPATHY (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 4
RENAL COLIC (Renal and urinary disorders) | 4
RENAL FAILURE (Renal and urinary disorders) | 1
URETHRAL DISORDER (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
BALANOPOSTHITIS (Reproductive system and breast disorders) | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 3
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 4
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 1
METRORRHAGIA (Reproductive system and breast disorders) | 1
UTERINE DISORDER (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
VULVAL ULCERATION (Reproductive system and breast disorders) | 1
VULVAR EROSION (Reproductive system and breast disorders) | 1
VULVOVAGINAL ERYTHEMA (Reproductive system and breast disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 12
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 11
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 1
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1
VOCAL CORD DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
ACNE (Skin and subcutaneous tissue disorders) | 6
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 7
ALOPECIA AREATA (Skin and subcutaneous tissue disorders) | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1
CHRONIC PIGMENTED PURPURA (Skin and subcutaneous tissue disorders) | 1
CUTANEOUS LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 1
DERMAL CYST (Skin and subcutaneous tissue disorders) | 2
DERMATITIS (Skin and subcutaneous tissue disorders) | 8
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 4
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 2
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 18
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 4
ECZEMA (Skin and subcutaneous tissue disorders) | 22
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 2
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 5
GRANULOMA SKIN (Skin and subcutaneous tissue disorders) | 1
GUTTATE PSORIASIS (Skin and subcutaneous tissue disorders) | 1
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 1
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 4
HYPERSENSITIVITY VASCULITIS (Skin and subcutaneous tissue disorders) | 2
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 1
LICHEN SCLEROSUS (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
PALMOPLANTAR KERATODERMA (Skin and subcutaneous tissue disorders) | 1
PRURIGO (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 11
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 3
PSORIASIS (Skin and subcutaneous tissue disorders) | 66
PURPURA (Skin and subcutaneous tissue disorders) | 1
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 21
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 2
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 1
ROSACEA (Skin and subcutaneous tissue disorders) | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 3
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 2
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 2
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 2
SKIN LESION (Skin and subcutaneous tissue disorders) | 7
SKIN MASS (Skin and subcutaneous tissue disorders) | 1
SKIN PLAQUE (Skin and subcutaneous tissue disorders) | 2
SKIN REACTION (Skin and subcutaneous tissue disorders) | 4
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2
TONSILLECTOMY (Surgical and medical procedures) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 9
VASCULITIS (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.